CLINICAL TRIAL: NCT04402450
Title: A Randomized Comparison Between Ultrasound-Guided Suprainguinal Fascia Iliaca Block and Pericapsular Nerve Group Block For Total Hip Replacement
Brief Title: Suprainguinal Fascia Iliaca Block Versus PENG Block for Hip Arthroplasty Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Julian Aliste, Assistant Professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: OAIC 1111/20
Record Dates: First submitted 2020-05-13; First posted 2020-05-26 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Complications; Postoperative Pain; Weakness, Muscle; Motor Activity
MeSH Terms: conditions — Postoperative Complications; Pain, Postoperative; Muscle Weakness; Motor Activity

STUDY DESIGN:
Intervention Model Description: prospective randomized comparison between two analgesic techniques
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- suprainguinal fascia iliaca block (Active Comparator): Forty mL of levobupivacaine 0.25% with epinephrine 5 ug/mL will be injected cranial to the inguinal ligament between the fascia iliaca and the iliopsoas muscle.
  Interventions: Procedure: Ultrasound-guided suprainguinal fascia iliaca nerve block
- Pericapsular nerve group block (Experimental): Twenty mL of levobupivacaine 0.5% with epinephrine 5 ug/mL will be deposited in the anterior aspect of the iliac bone between its periosteum and the tendon of the iliopsoas muscle.
  Interventions: Procedure: Ultrasound-guided pericapsular nerves group of the hip block

INTERVENTIONS:
Procedure: Ultrasound-guided suprainguinal fascia iliaca nerve block — After an ultrasound-guided insertion of a block needle below the inguinal ligament, the needle will be advance in the plane between fascia iliaca and iliopsoas muscle up to a point cranial to the ligament in order to inject a 40 mL of adrenalized 0.25% levobupivacaine.
  Arms: suprainguinal fascia iliaca block
Procedure: Ultrasound-guided pericapsular nerves group of the hip block — After an ultrasound-guided insertion of a block needle at the level of the inguinal ligament, the needle will be advance into the plane between iliac bone periosteum and the tendon of the iliopsoas muscle in order to inject 20 mL of adrenalized 0.5% levobupivacaine.
  Arms: Pericapsular nerve group block

SUMMARY:
In recent years, suprainguinal fascia iliaca block (SFIB) has emerged as a reliable analgesic option for primary total hip arthroplasty (THA). In 2018, a new block was described, termed pericapsular nerve group block or PENG block, that selectively targets the articular branches of the femoral and obturator nerves while sparing their motor components. In this randomized trial, the investigators will compare US-guided SFIB and PENG block in patients undergoing primary THA. Since the main benefit of PENGB stems from its quadriceps-sparing effect, it was selected the incidence of quadriceps motor block (at 6 hours) as the primary outcome and the hypothesis that PENG block will result in significantly less motor block compared to SFIB.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* American Society of Anesthesiologists classification 1-3
* Body mass index between 20 and 35 (kg/m2)

Exclusion Criteria:

* Adults who are unable to give their own consent
* Pre-existing neuropathy (assessed by history and physical examination)
* Coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. platelets ≤a100, International Normalized Ratio ≥01.4 or prothrombin time ≥ 50)
* Renal failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. creatinine ≥ 100)
* Hepatic failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. transaminases ≥ 100)
* Allergy to local anesthetics (LAs)
* Pregnancy
* Prior surgery in the corresponding side of the inguinal or suprainguinal area
* Chronic pain syndromes requiring opioid intake at home

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Presence of quadriceps motor block (defined as paralysis or paresis). | 6 hours after block performance
  Quadriceps motor function will be tested with the patient supine and with the hip and knee flexed at 45º and 90º, respectively. The subject will be asked to extend the knee first against gravity and then against resistance. Quadriceps strength will be graded according to a 3-point scale: normal strength = 0 point (extension against resistance); paresis = 1 point (extension against gravity but not against resistance); and paralysis = 2 points (no extension).

SECONDARY OUTCOMES:
Block performance time | 1 hour after surgery
  temporal interval between the start of skin disinfection and the end of LA injection through the block needle
Static and dynamic pain | 3 hours after the block
  Pain intensity at rest and during active movement using a numeric rating score (NRS) ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Static and dynamic pain | 6 hours after the block
  Pain intensity at rest and during active movement using a numeric rating score (NRS) ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Static and dynamic pain | 12 hours after the block
  Pain intensity at rest and during active movement using a numeric rating score (NRS) ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Static and dynamic pain | 18 hours after the block
  Pain intensity at rest and during active movement using a numeric rating score (NRS) ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Static and dynamic pain | 24 hours after the block
  Pain intensity at rest and during active movement using a numeric rating score (NRS) ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Static and dynamic pain | 36 hours after the block
  Pain intensity at rest and during active movement using a numeric rating score (NRS) ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Static and dynamic pain | 48 hours after the block
  Pain intensity at rest and during active movement using a numeric rating score (NRS) ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Postoperative morphine consumption | 24 hours after the block
  consumption of intravenous morphine registered by a patient controlled analgesia device
Postoperative morphine consumption | 48 hours after the block
  consumption of intravenous morphine registered by a patient controlled analgesia device
Sensory block | 3 hours after the block
  Sensory block in the anterior, lateral and medial aspects of the mid-thigh. For each territory, blockade will be evaluated using a 3-point scale: 0 = no block, 1 = analgesia (patient can feel touch, not cold), 2 = anesthesia (patient cannot feel touch)
Sensory block | 6 hours after the block
  Sensory block in the anterior, lateral and medial aspects of the mid-thigh. For each territory, blockade will be evaluated using a 3-point scale: 0 = no block, 1 = analgesia (patient can feel touch, not cold), 2 = anesthesia (patient cannot feel touch)
Sensory block | 24 hours after the block
  Sensory block in the anterior, lateral and medial aspects of the mid-thigh. For each territory, blockade will be evaluated using a 3-point scale: 0 = no block, 1 = analgesia (patient can feel touch, not cold), 2 = anesthesia (patient cannot feel touch)
Presence of quadriceps motor block (defined as paralysis or paresis). | 3 hours after the block
  Quadriceps motor function will be tested with the patient supine and with the hip and knee flexed at 45º and 90º, respectively. The subject will be asked to extend the knee first against gravity and then against resistance. Quadriceps strength will be graded according to a 3-point scale: normal strength = 0 point (extension against resistance); paresis = 1 point (extension against gravity but not against resistance); and paralysis = 2 points (no extension).
Presence of quadriceps motor block (defined as paralysis or paresis). | 24 hours after the block
  Quadriceps motor function will be tested with the patient supine and with the hip and knee flexed at 45º and 90º, respectively. The subject will be asked to extend the knee first against gravity and then against resistance. Quadriceps strength will be graded according to a 3-point scale: normal strength = 0 point (extension against resistance); paresis = 1 point (extension against gravity but not against resistance); and paralysis = 2 points (no extension).
Hip adduction strength. | 3 hours after the block
  Hip adduction will be evaluated by comparing it to baseline strength (i.e., prior to spinal anesthesia). A blood pressure cuff, inflated at 40 mmHg, will be inserted between the knees of the patient: the latter will then be instructed to squeeze the cuff as hard as possible and to sustain the effort. We will define hip adduction scores of 0, 1 and 2 points as decreases in strength of 0-20%, 21-70% and 71-90% compared to baseline measurement, respectively.
Hip adduction strength. | 6 hours after the block
  Hip adduction will be evaluated by comparing it to baseline strength (i.e., prior to spinal anesthesia). A blood pressure cuff, inflated at 40 mmHg, will be inserted between the knees of the patient: the latter will then be instructed to squeeze the cuff as hard as possible and to sustain the effort. We will define hip adduction scores of 0, 1 and 2 points as decreases in strength of 0-20%, 21-70% and 71-90% compared to baseline measurement, respectively.
Hip adduction strength. | 24 hours after the block
  Hip adduction will be evaluated by comparing it to baseline strength (i.e., prior to spinal anesthesia). A blood pressure cuff, inflated at 40 mmHg, will be inserted between the knees of the patient: the latter will then be instructed to squeeze the cuff as hard as possible and to sustain the effort. We will define hip adduction scores of 0, 1 and 2 points as decreases in strength of 0-20%, 21-70% and 71-90% compared to baseline measurement, respectively.
Block-related complications | 1 hour after the block
  vascular puncture, paresthesia or systemic local anesthetic toxicity
Postoperative opioid related side effects | 48 hours after the block
  Presence of postoperative nausea, vomiting, pruritus, urinary retention, respiratory depression
Inability to perform physiotherapy due to motor block | Postoperative day 1
  Number of participants that cannot end the physiotherapy protocol programmed for the first postoperative day secondary to decreased strength in the operated leg.
Inability to perform physiotherapy due to motor block | postoperative day 2
  Number of participants that cannot end the physiotherapy protocol programmed for the second postoperative day secondary to decreased strength in the operated leg.
Inability to perform physiotherapy due to pain | postoperative day 1
  Number of participants that cannot end the physiotherapy protocol programmed for the first postoperative day secondary to pain in the operated leg.
Inability to perform physiotherapy due to pain | postoperative day 2
  Number of participants that cannot end the physiotherapy protocol programmed for the second postoperative day secondary to pain in the operated leg.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universidad de Chile, Santiago, Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No
unidentified data can be shared upon reasonable request after study publication

REFERENCES:
- [Result] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Result] Hebbard P, Ivanusic J, Sha S. Ultrasound-guided supra-inguinal fascia iliaca block: a cadaveric evaluation of a novel approach. Anaesthesia. 2011 Apr;66(4):300-5. doi: 10.1111/j.1365-2044.2011.06628.x. Epub 2011 Feb 24. PMID 21401544
- [Derived] Aliste J, Layera S, Bravo D, Jara A, Munoz G, Barrientos C, Wulf R, Branez J, Finlayson RJ, Tran Q. Randomized comparison between pericapsular nerve group (PENG) block and suprainguinal fascia iliaca block for total hip arthroplasty. Reg Anesth Pain Med. 2021 Oct;46(10):874-878. doi: 10.1136/rapm-2021-102997. Epub 2021 Jul 20. PMID 34290085